CLINICAL TRIAL: NCT07404631
Title: Effect of Intermittent Pneumatic Compression on Ankle Joint Proprioception and Balance in Patients With Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ashraf Sayed Abd El Hadi, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005794
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermitted pneumatic pressure + Conventional physical therapy (Experimental): Participants will receive the intermitted pneumatic pressure in addition to conventional physical therapy, 3 times per week for six weeks.
  Interventions: Device: Intermitted pneumatic pressure; Other: Conventional physical therapy
- Conventional physical therapy (Active Comparator): Participants will receive conventional physical therapy only, 3 times per week for six weeks.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Intermitted pneumatic pressure — Intermittent pneumatic compression will be applied with the patient positioned comfortably in a supported supine lying position on an appropriately sized treatment table. The treated limb will be inspected for skin integrity, with any bandages removed, and a cotton gauze sleeve will be applied prior to placement of the compression sleeve. The compression unit will be placed on a stable surface, checked for cleanliness and proper assembly, and securely connected to the limb. Treatment parameters will be set at a pressure of 40 mmHg with an intermittent cycle of 90 seconds of inflation followed by 90 seconds of deflation. Each treatment session will last 30 minutes.
  Arms: Intermitted pneumatic pressure + Conventional physical therapy
Other: Conventional physical therapy — Conventional physical therapy will be received in the form of range of motion exercises, strength exercise, stretching exercises, sit to stand, proprioception training and balance training, 3 times per week for 6 weeks.

SUMMARY:
This study aims to assess the effect of intermittent pneumatic compression on ankle joint proprioception and balance in patients with stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability worldwide, often resulting in motor impairments that limit mobility, daily activities, social participation, and overall quality of life. Although many stroke survivors regain independent ambulation, deficits in balance, posture, and gait commonly persist due to impaired voluntary motor control of the paretic lower limb. Recovery of lower limb motor function is essential for walking, independence in activities of daily living, and social participation. Proprioception, which provides sensory information about body position and movement, plays a critical role in motor control and functional performance. Proprioceptive deficits are common after stroke and are more pronounced in the lower limb, contributing to impaired balance, gait disturbances, and increased fall risk. Stroke rehabilitation aims to restore function through interventions that enhance sensory input, promote cortical plasticity, and improve motor recovery. Therefore, this study aims to assess the effect of intermittent pneumatic compression on ankle joint proprioception and balance in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patients will range from 50-65 years old.
* Patients with stroke duration of illness ranged from six months to 18 months.
* BMI (Body Mass Index) ranged from 20- 30 Kg/m2.
* The muscle tone of the affected lower limb muscles ranged from 1 to 2 grade according Modified Aschworth Scale.
* Patients who have moderate impaired balance.
* Patients who have impaired proprioception.

Exclusion Criteria:

* Patients with cardiovascular problems (open heart surgery or pacemaker).
* Patients with neurological diseases that affect lower limb function other than stroke (ex: Multiple sclerosis, Peripheral neuropathy, Parkinsonism…. etc.).
* Patients Suffered of Deep veins thrombosis (DVT).
* Patient with recurrent stroke.
* Patients with musculoskeletal disorders such as severe arthritis, knee surgery, total hip joint replacement, lower limb fractures or contractures of fixed deformity, leg length discrepancy after total hip replacement

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
Ankle proprioception | 6 weeks
  It will be assessed by measuring the absolute error between target and reproduced ankle angles using an isokinetic dynamometer. Participants attempt to reproduce 10° and 20° of plantar flexion without visual feedback. The absolute error represents the difference between the target and reproduced angles. Smaller errors indicate better proprioceptive accuracy, while larger errors reflect impaired proprioception.
Mediolateral Stability Index (MLSI) | 6 weeks
  It reflects the individual's ability to control balance from side to side. Measured on the Biodex Balance System, it quantifies mediolateral sway. Higher MLSI values indicate increased instability, while lower values reflect better control. It is particularly useful for assessing balance deficits in conditions like stroke, where lateral stability is often impaired, aiding in targeted rehabilitation strategies.
Anteroposterior Stability Index (APSI) | 6 weeks
  It measures front-to-back balance control using the Biodex Balance System. It evaluates how well an individual stabilizes posture in the forward and backward directions. Elevated APSI scores indicate greater postural sway and instability, while lower scores indicate better balance. This index is critical in identifying anteroposterior balance deficits and guiding targeted rehabilitation.
Overall Stability Index (OSI) | 6 weeks
  is a composite measure reflecting balance control in all directions-mediolateral and anteroposterior. Assessed via the Biodex Balance System, a higher OSI indicates greater overall body sway and instability. Lower OSI values reflect better multi-directional balance. This index is crucial in providing a global assessment of postural control and is used to monitor progress in balance rehabilitation.

SECONDARY OUTCOMES:
Limits of Stability (LOS) score | 6 weeks
  LOS test evaluates patient's ability to intentionally shift center of gravity in eight directions (Forward, Backward, Right, Left, Forward-Right, Forward-Left, Backward-Right, Backward-Left) without losing balance. Three trials per direction; averages calculated. Lower scores indicate restricted stability limits common post-stroke, affecting functional mobility and fall risk.
The Berg Balance Scale (BBS) | 6 weeks
  It is a 14-item clinical test used to objectively measure balance ability during functional tasks. Each task is scored from 0 (unable) to 4 (independent), with a total score out of 56. Lower scores indicate higher fall risk. It assesses static and dynamic balance in tasks like standing, turning, and reaching. The BBS is widely used in stroke rehabilitation to evaluate balance improvements over time.
The Timed Up and Go (TUG) test | 6 weeks
  It measures functional mobility and fall risk. Participants stand from a chair, walk 3 meters, turn, return, and sit. The time in seconds is recorded. A completion time of ≥12 seconds indicates increased fall risk. The TUG is a simple, reliable test used in clinical settings to track progress in mobility and balance rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Sadik Badway, PhD, Study Chair — Professor, Cairo University; Ebtessam Mohamed Fahmy, PhD, Study Director — Professor, Cairo University; Nagwa Ibrahim Rehab, PhD, Study Director — Assis. Professor, Cairo University
Locations (1):
- Ministry of Health, Cairo, Egypt